CLINICAL TRIAL: NCT03156127
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Study to Compare the Pharmacokinetics and Safety/Tolerability of BR-UPS (Ulipristal Acetate) 5 mg Tablet With Inisia (Ulipristal Acetate) 5 mg Tablet in Healthy Female Volunteers
Brief Title: A Study to Compare the Pharmacokinetics and Safety/Tolerability of BR-UPS (Ulipristal Acetate) 5 mg Tablet With Inisia (Ulipristal Acetate) 5 mg Tablet
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Problem of Investigational Products
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-UPS-CT-101
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Uterine Myoma
MeSH Terms: conditions — Myofibroma | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR-UPS 5 mg tablet (Experimental)
  Interventions: Drug: BR-UPS 5 mg tablet, Inisia 5 mg tablet
- Inisia 5 mg tablet (Active Comparator)
  Interventions: Drug: BR-UPS 5 mg tablet, Inisia 5 mg tablet

INTERVENTIONS:
Drug: BR-UPS 5 mg tablet, Inisia 5 mg tablet — Subjects of Control group will be first orally administered with inisia 5mg tablet . After washout period of 2 weeks, They will be orally administered with BR-UPS 5mg tablet. On the contrary, Subjects of Test group will be first orally administered with BR-UPS 5mg tablet. After washout period of 2 weeks, They will be orally administered with inisia 5mg tablet.

SUMMARY:
The purpose of this study is to evaluate the Pharmacokinetics and Safety / Tolerability of BR-UPS (Ulipristal acetate) 5 mg tablet with Inisia (Ulipristal acetate) 5 mg tablet in healthy female volunteers

DETAILED DESCRIPTION:
This is a randomized, open-label, single dose, two-way crossover study to compare the pharmacokinetics and safety/tolerability of BR-UPS (Ulipristal acetate) 5 mg tablet with Inisia (Ulipristal acetate) 5 mg tablet in healthy female volunteers

ELIGIBILITY:
Inclusion Criteria:

* A subject provide written informed consent which he voluntarily confirms willingness to participate in a study, having been informed of the full details of the study and comply with the protocol.
* A Healthy female volunteers, aged 19-45 years
* BMI 18 ~ 27(kg/m2)

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease.
* History of gastrointestinal disease and resection
* History of clinically significant hypersensitivity to study drug, any other drug
* A subject with clinically significant genital bleeding
* Participation in any other study within 3 months
* Positive results for urine β-hCG in screening or lactating women
* A subject is using a method of hormone contraception and a Progesterone intrauterine device

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Cmax(Maximum concentration of drug in plasma) of Ulipristal Acetate | 0~120 hours after medication
AUClast(Area under the plasma drug concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration) of Ulipristal Acetate | 0~120 hours after medication

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No